CLINICAL TRIAL: NCT03412383
Title: A Phase II Study of Pyrotinib in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer
Brief Title: Pyrotinib in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Clinical Professor, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201711008
Record Dates: First submitted 2018-01-14; First posted 2018-01-26 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; HER2 Gene Mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400mg/day

SUMMARY:
A Phase II Study of Pyrotinib in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

Able to understand and willing to sign an Institutional Review Board（IRB） approved written informed consent document.

At least 18 years of age. Histologically or cytologically confirmed HER2-negative (0 or 1+ by immuno-histochemical (IHC) or non-amplified by FISH) breast cancer that is stage IV.

There is no standard therapy. At least one measurable disease by RECIST 1.1 is required. Karnofsky performance status (KPS)>70, life expectancy > 12 weeks

Exclusion Criteria:

Lack of adequate organ function as defined below within 2 weeks of registration:

Absolute neutrophil count (ANC)<1.5×109/L，platelet counts (PLT)<75×109/L or hemoglobin (Hb)<100g/L Total bilirubin (TBiL)>2×upper limit of normal (ULN); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>2.5×ULN（or>5 x ULN for patients with liver metastases）; Alkaline phosphatase (ALP)>2.5×ULN; serum creatinine concentration (Scr)>140umol/L Pregnant and/or breastfeeding. History of significant cardiac disease, cardiac risk factors, or uncontrolled arrhythmias.

Having a history of uncontrolled paroxysmal diseases, including central nervous system diseases or mental disorders which may have an impact on the understanding and signature of informed consent Uncontrolled acute infection Currently receiving any other investigational agents or systemic cancer therapy.

Allergy to any investigational drug ; Any other condition that investigator considers inappropriate to participate in this trail

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-02-20 (Estimated); Primary Completion 2019-01-25 (Estimated); Study Completion 2019-06-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 36 months
  From date of first use Pyrotinib until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Adverse events (AEs) | up to 36 months
  Adverse events (AEs) and laboratory tests graded according to the NCI CTCAE (version 4.0)
Overall Response rates (ORR) | up to 36 months
  Defined as complete response (CR) + partial response (PR), assessed based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria.
Clinical Benefit rate (CBR) | up to 36 months
  Defined as CR+PR+stable disease (SD), assessed based on on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria.
Time to Progression (TTP) | up to 36 months
  Time from first use Pyrotinib to disease progression
Quality of Life(QoL) | up to 36 months
  Using the EORTC quality of life questionnaire QLQ-C30
Overall survival (OS) | up to 52 months
  Time from first use Pyrotinib to death

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Fei Ma, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yi Z, Feng K, Lv D, Guan Y, Shao Y, Ma F, Xu B. Genomic landscape of circulating tumor DNA in HER2-low metastatic breast cancer. Signal Transduct Target Ther. 2024 Dec 9;9(1):345. doi: 10.1038/s41392-024-02047-0. PMID 39648226